CLINICAL TRIAL: NCT03461432
Title: Testing the Feasibility and Acceptability of a New Personalised Form of Cognitive Remediation Therapy (pCRT) for People With Psychosis.
Brief Title: Personalised Cognitive Remediation Therapy (pCRT)
Acronym: pCRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 231245
Record Dates: First submitted 2018-02-15; First posted 2018-03-12 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-02

CONDITIONS: Schizophrenia Schizoaffective
Keywords: Cognitive Remediation Therapy CRT
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: A case-control study design with pre- and post-therapy assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalised Cognitive Remediation Therapy (pCRT) (Experimental): A case-control study design with pre- and post-therapy assessment, comparing a group of participants with schizophrenia who received standard CRT, with a similar group of participants receiving pCRT.
  Interventions: Behavioral: Cognitive Remediation Therapy

INTERVENTIONS:
Behavioral: Cognitive Remediation Therapy — Cognitive Remediation Therapy (CRT) is a psychological therapy that has been developed with a general immediate focus on improving impaired cognitive domains but ultimately aimed at improving social and functional outcomes.

SUMMARY:
Cognitive deficits have been shown to have negative impact on social functioning and functional goals such as ability to work and perform daily tasks in people with schizophrenia. There is evidence that Cognitive Remediation Therapy, a form of psychological therapy, is effective in improving cognition and functioning but there is still a limited understanding of what influence people's different response to this therapy. A tailored treatment is likely to be more effective because it will adapt to service users' unique characteristics.

The investigators are planning a study exploring at the feasibility and acceptability of novel form of Cognitive Remediation Therapy which is personalised (pCRT) to the person individual characteristics. The personalised therapy will consist of task practice using computerized Cognitive Remediation software (i.e. called CIRCuiTS). The knowledge gathered in this work will contribute to develop the next generation of personalised treatment approaches for people with schizophrenia.

DETAILED DESCRIPTION:
Cognitive deficits in people with psychosis have been shown to have negative impact on functional goals including the ability to work and perform daily tasks. Cognitive Remediation Therapy (CRT) is a psychological therapy developed to improve cognitive functions in people with schizophrenia but ultimately with a focus on improving social and functional outcomes. There is evidence that CRT is effective in improving cognition and functioning but there is still a limited understanding of the mechanisms responsible for different treatment responses. This study attempts to fill this gap by developing and testing a new form of CRT, which will personalise therapy elements according to participants' characteristics. The therapy will consist of task practice using a computerised Cognitive Remediation software and supervised activities supported by a therapist to boost functioning. The knowledge gathered in this work will contribute to develop the next generation of personalised treatment approaches for people with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* a range of 18-65 years
* English speaking or with a good knowledge of the language
* a diagnosis of schizophrenia or schizoaffective disorder according to the DSM- V
* at least one year contact with mental health services,
* a deficit (of at least one standard deviation below the mean) in at least one cognitive domain out of these three cognitive domains: memory, executive function and information processing.

Exclusion Criteria:

* Planned medication change
* Diagnosis of learning disability
* Presence of cognitive deficits related to organic causes or head injury
* Primary diagnosis of substance dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-10-31 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of intervention (including acceptance rates, drop outs) | 3 months post baseline assessment
  Feasibility estimates of delivering the intervention including acceptance rates, drop outs.

SECONDARY OUTCOMES:
Acceptability of intervention (Satisfaction) | 3 months post baseline assessment
  Questionnaire of Satisfaction

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wykes T, Huddy V, Cellard C, McGurk SR, Czobor P. A meta-analysis of cognitive remediation for schizophrenia: methodology and effect sizes. Am J Psychiatry. 2011 May;168(5):472-85. doi: 10.1176/appi.ajp.2010.10060855. Epub 2011 Mar 15. PMID 21406461